CLINICAL TRIAL: NCT02921321
Title: Pilot Study of Cardiac Magnetic Resonance in Patients With Muscular Dystrophy
Brief Title: Pilot Study of Cardiac MR in Patients With Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Christopher Spurney, MD, Children's National Research Institute
Other Study IDs: 4193; Internal Bridge Funding (Other: Children's Research Institute,Children's National)
Record Dates: First submitted 2016-08-29; First posted 2016-10-03 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Muscular Dystrophies; Cardiac Fibrosis; Genetic Diseases, Inborn; Musculoskeletal Diseases
Keywords: MRI; Muscular Dystrophy; Cardiac; Late gadolinium enhancement
MeSH Terms: conditions — Muscular Dystrophies; Genetic Diseases, Inborn; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An additional 5cc of blood work will be drawn at the time that the intravascular catheter is inserted for contrast agent administration for the cardiac MRI scans. This blood will be used to identify serum biomarkers in myocardial fibrosis, and to validate the potential use for diagnostic purposes. No genetic testing will be done on these samples. The blood samples will be identified with the study ID number only, and will be stored in a secure freezer.
Oversight: Data Monitoring Committee: No

SUMMARY:
Muscular Dystrophy can affect the skeletal muscles and also the heart and breathing muscles, causing significant morbidity and mortality. As patients are now living longer, treatment of muscular dystrophies involves drugs that help improve heart function. However, better types of heart imaging studies are needed to understand how these treatments work. Researchers want to improve heart imaging to identify earlier indicators of heart dysfunction in muscular dystrophy patients and how these are changed by medical treatment. The new imaging indicators will also help identify candidates for entry into future clinical trials.

DETAILED DESCRIPTION:
Cardiomyopathy causes significant morbidity and mortality in multiple forms of muscular dystrophy affecting children, including Duchenne muscular dystrophy (DMD), Becker muscular dystrophy (BMD) and subtypes of autosomal recessive limb-girdle muscular dystrophy (LGMD2). Pharmaceutical treatments for the cardiomyopathy of muscular dystrophy, including angiotensin-converting enzyme (ACE) inhibition and beta-adrenergic receptor blockade, afford significant benefit and demonstrate cardiac remodeling in clinical studies. Further studies are needed to identify and characterize more sensitive indicators of cardiac dysfunction in muscular dystrophy subjects to better stratify subjects for entry into clinical protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Duchenne, Becker, or Limb Girdle Muscular Dystrophy

Exclusion Criteria:

* Day-time users of continuous positive airway pressure (CPAP)
* Sip ventilator users
* Invasive ventilator dependent
* Pregnant minors or adults (when uncertain, participants will undergo urine testing) or lactating minors and adults
* Females who are nursing and who do not plan to discard breast milk for 24 hours
* Decompensated congestive heart failure (unable to lie flat during CMR)
* Impaired renal excretory function (calculated Glomerular Filtration Rate less than 30 milliliters/min)
* Contra-indications to Magnetic Resonance Imaging:
* Cardiac pacemaker or implantable defibrillator
* Cerebral aneurysm clip
* Neural stimulator
* Metallic ocular foreign body
* Any implanted device (i.e. insulin pump, drug infusion device)
* Claustrophobia
* Metal shrapnel or bullet
* Investigator assessment of inability to comply with protocol
* Unable/unwilling to lie still throughout the research procedure or who require sedation
* Persons with cognitive impairment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or females at least 6 years of age with a diagnosis of Duchenne, Becker, or Limb Girdle Muscular Dystrophy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Myocardial characterization of fibrosis in patients with muscular dystrophy using contrast based magnetic resonance imaging | At the end of each MRI scan through study completion, up to 5 years.

SECONDARY OUTCOMES:
Measure the amount of intramyocardial fibrosis using extracellular volume measurements | At the end of each MRI scan through study completion, up to 5 years.
Identification and validation of serum biomarker ST2 (Interleukin 1 receptor-like 1 protein ) in the presence of myocardial fibrosis. | At the end of the study, up to 10 years
Measure regional myocardial strain and correlate with presence of myocardial fibrosis | At the end of each MRI scan through study completion, up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Spurney, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman EP, Brown RH Jr, Kunkel LM. Dystrophin: the protein product of the Duchenne muscular dystrophy locus. Cell. 1987 Dec 24;51(6):919-28. doi: 10.1016/0092-8674(87)90579-4. PMID 3319190
- [Background] Nigro G, Comi LI, Politano L, Bain RJ. The incidence and evolution of cardiomyopathy in Duchenne muscular dystrophy. Int J Cardiol. 1990 Mar;26(3):271-7. doi: 10.1016/0167-5273(90)90082-g. PMID 2312196
- [Background] Corrado G, Lissoni A, Beretta S, Terenghi L, Tadeo G, Foglia-Manzillo G, Tagliagambe LM, Spata M, Santarone M. Prognostic value of electrocardiograms, ventricular late potentials, ventricular arrhythmias, and left ventricular systolic dysfunction in patients with Duchenne muscular dystrophy. Am J Cardiol. 2002 Apr 1;89(7):838-41. doi: 10.1016/s0002-9149(02)02195-1. PMID 11909570
- [Background] Mendell JR, Moxley RT, Griggs RC, Brooke MH, Fenichel GM, Miller JP, King W, Signore L, Pandya S, Florence J, et al. Randomized, double-blind six-month trial of prednisone in Duchenne's muscular dystrophy. N Engl J Med. 1989 Jun 15;320(24):1592-7. doi: 10.1056/NEJM198906153202405. PMID 2657428
- [Background] Cox GF, Kunkel LM. Dystrophies and heart disease. Curr Opin Cardiol. 1997 May;12(3):329-43. PMID 9243091
- [Background] Deburgrave N, Daoud F, Llense S, Barbot JC, Recan D, Peccate C, Burghes AH, Beroud C, Garcia L, Kaplan JC, Chelly J, Leturcq F. Protein- and mRNA-based phenotype-genotype correlations in DMD/BMD with point mutations and molecular basis for BMD with nonsense and frameshift mutations in the DMD gene. Hum Mutat. 2007 Feb;28(2):183-95. doi: 10.1002/humu.20422. PMID 17041906
- [Background] Mathews KD, Moore SA. Limb-girdle muscular dystrophy. Curr Neurol Neurosci Rep. 2003 Jan;3(1):78-85. doi: 10.1007/s11910-003-0042-9. PMID 12507416
- [Background] Lim LE, Campbell KP. The sarcoglycan complex in limb-girdle muscular dystrophy. Curr Opin Neurol. 1998 Oct;11(5):443-52. doi: 10.1097/00019052-199810000-00006. PMID 9847993
- [Background] Turakhia MP, Schiller NB, Whooley MA. Prognostic significance of increased left ventricular mass index to mortality and sudden death in patients with stable coronary heart disease (from the Heart and Soul Study). Am J Cardiol. 2008 Nov 1;102(9):1131-5. doi: 10.1016/j.amjcard.2008.06.036. Epub 2008 Aug 27. PMID 18940278
- [Background] Devereux RB, Lutas EM, Casale PN, Kligfield P, Eisenberg RR, Hammond IW, Miller DH, Reis G, Alderman MH, Laragh JH. Standardization of M-mode echocardiographic left ventricular anatomic measurements. J Am Coll Cardiol. 1984 Dec;4(6):1222-30. doi: 10.1016/s0735-1097(84)80141-2. PMID 6238987
- [Background] Gardin JM, McClelland R, Kitzman D, Lima JA, Bommer W, Klopfenstein HS, Wong ND, Smith VE, Gottdiener J. M-mode echocardiographic predictors of six- to seven-year incidence of coronary heart disease, stroke, congestive heart failure, and mortality in an elderly cohort (the Cardiovascular Health Study). Am J Cardiol. 2001 May 1;87(9):1051-7. doi: 10.1016/s0002-9149(01)01460-6. PMID 11348601
- [Background] Haider AW, Larson MG, Benjamin EJ, Levy D. Increased left ventricular mass and hypertrophy are associated with increased risk for sudden death. J Am Coll Cardiol. 1998 Nov;32(5):1454-9. doi: 10.1016/s0735-1097(98)00407-0. PMID 9809962
- [Background] Lavie CJ, Milani RV, Ventura HO, Messerli FH. Left ventricular geometry and mortality in patients >70 years of age with normal ejection fraction. Am J Cardiol. 2006 Nov 15;98(10):1396-9. doi: 10.1016/j.amjcard.2006.06.037. Epub 2006 Oct 2. PMID 17134637
- [Background] Verdecchia P, Carini G, Circo A, Dovellini E, Giovannini E, Lombardo M, Solinas P, Gorini M, Maggioni AP; MAVI (MAssa Ventricolare sinistra nell'Ipertensione) Study Group. Left ventricular mass and cardiovascular morbidity in essential hypertension: the MAVI study. J Am Coll Cardiol. 2001 Dec;38(7):1829-35. doi: 10.1016/s0735-1097(01)01663-1. PMID 11738281
- [Background] Bluemke DA, Kronmal RA, Lima JA, Liu K, Olson J, Burke GL, Folsom AR. The relationship of left ventricular mass and geometry to incident cardiovascular events: the MESA (Multi-Ethnic Study of Atherosclerosis) study. J Am Coll Cardiol. 2008 Dec 16;52(25):2148-55. doi: 10.1016/j.jacc.2008.09.014. PMID 19095132
- [Background] Kannel WB, Gordon T, Castelli WP, Margolis JR. Electrocardiographic left ventricular hypertrophy and risk of coronary heart disease. The Framingham study. Ann Intern Med. 1970 Jun;72(6):813-22. doi: 10.7326/0003-4819-72-6-813. No abstract available. PMID 4247338
- [Background] Levy D, Garrison RJ, Savage DD, Kannel WB, Castelli WP. Left ventricular mass and incidence of coronary heart disease in an elderly cohort. The Framingham Heart Study. Ann Intern Med. 1989 Jan 15;110(2):101-7. doi: 10.7326/0003-4819-110-2-101. PMID 2521199
- [Background] Levy D, Garrison RJ, Savage DD, Kannel WB, Castelli WP. Prognostic implications of echocardiographically determined left ventricular mass in the Framingham Heart Study. N Engl J Med. 1990 May 31;322(22):1561-6. doi: 10.1056/NEJM199005313222203. PMID 2139921
- [Background] Devereux RB, Dahlof B, Gerdts E, Boman K, Nieminen MS, Papademetriou V, Rokkedal J, Harris KE, Edelman JM, Wachtell K. Regression of hypertensive left ventricular hypertrophy by losartan compared with atenolol: the Losartan Intervention for Endpoint Reduction in Hypertension (LIFE) trial. Circulation. 2004 Sep 14;110(11):1456-62. doi: 10.1161/01.CIR.0000141573.44737.5A. Epub 2004 Aug 23. PMID 15326072
- [Background] Devereux RB, Wachtell K, Gerdts E, Boman K, Nieminen MS, Papademetriou V, Rokkedal J, Harris K, Aurup P, Dahlof B. Prognostic significance of left ventricular mass change during treatment of hypertension. JAMA. 2004 Nov 17;292(19):2350-6. doi: 10.1001/jama.292.19.2350. PMID 15547162
- [Background] Kjeldsen SE, Dahlof B, Devereux RB, Julius S, Aurup P, Edelman J, Beevers G, de Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Snapinn S, Wedel H; LIFE (Losartan Intervention for Endpoint Reduction) Study Group. Effects of losartan on cardiovascular morbidity and mortality in patients with isolated systolic hypertension and left ventricular hypertrophy: a Losartan Intervention for Endpoint Reduction (LIFE) substudy. JAMA. 2002 Sep 25;288(12):1491-8. doi: 10.1001/jama.288.12.1491. PMID 12243636
- [Background] Okin PM, Devereux RB, Jern S, Kjeldsen SE, Julius S, Nieminen MS, Snapinn S, Harris KE, Aurup P, Edelman JM, Wedel H, Lindholm LH, Dahlof B; LIFE Study Investigators. Regression of electrocardiographic left ventricular hypertrophy during antihypertensive treatment and the prediction of major cardiovascular events. JAMA. 2004 Nov 17;292(19):2343-9. doi: 10.1001/jama.292.19.2343. PMID 15547161
- [Background] Bottini PB, Carr AA, Prisant LM, Flickinger FW, Allison JD, Gottdiener JS. Magnetic resonance imaging compared to echocardiography to assess left ventricular mass in the hypertensive patient. Am J Hypertens. 1995 Mar;8(3):221-8. doi: 10.1016/0895-7061(94)00178-E. PMID 7794570
- [Background] Caiani EG, Corsi C, Sugeng L, MacEneaney P, Weinert L, Mor-Avi V, Lang RM. Improved quantification of left ventricular mass based on endocardial and epicardial surface detection with real time three dimensional echocardiography. Heart. 2006 Feb;92(2):213-9. doi: 10.1136/hrt.2005.060889. Epub 2005 May 12. PMID 15890763
- [Background] Hees PS, Fleg JL, Lakatta EG, Shapiro EP. Left ventricular remodeling with age in normal men versus women: novel insights using three-dimensional magnetic resonance imaging. Am J Cardiol. 2002 Dec 1;90(11):1231-6. doi: 10.1016/s0002-9149(02)02840-0. PMID 12450604
- [Background] Solomon SD, Appelbaum E, Manning WJ, Verma A, Berglund T, Lukashevich V, Cherif Papst C, Smith BA, Dahlof B; Aliskiren in Left Ventricular Hypertrophy (ALLAY) Trial Investigators. Effect of the direct Renin inhibitor aliskiren, the Angiotensin receptor blocker losartan, or both on left ventricular mass in patients with hypertension and left ventricular hypertrophy. Circulation. 2009 Feb 3;119(4):530-7. doi: 10.1161/CIRCULATIONAHA.108.826214. Epub 2009 Jan 19. PMID 19153265
- [Background] de Lemos JA, McGuire DK, Khera A, Das SR, Murphy SA, Omland T, Drazner MH. Screening the population for left ventricular hypertrophy and left ventricular systolic dysfunction using natriuretic peptides: results from the Dallas Heart Study. Am Heart J. 2009 Apr;157(4):746-53.e2. doi: 10.1016/j.ahj.2008.12.017. Epub 2009 Feb 20. PMID 19332205
- [Background] Flacke SJ, Fischer SE, Lorenz CH. Measurement of the gadopentetate dimeglumine partition coefficient in human myocardium in vivo: normal distribution and elevation in acute and chronic infarction. Radiology. 2001 Mar;218(3):703-10. doi: 10.1148/radiology.218.3.r01fe18703. PMID 11230643
- [Background] Wu YL, Ye Q, Sato K, Foley LM, Hitchens TK, Ho C. Noninvasive evaluation of cardiac allograft rejection by cellular and functional cardiac magnetic resonance. JACC Cardiovasc Imaging. 2009 Jun;2(6):731-41. doi: 10.1016/j.jcmg.2009.01.013. PMID 19520344
- [Background] Harris PA, Lorenz CH, Holburn GE, Overholser KA. Regional measurement of the Gd-DTPA tissue partition coefficient in canine myocardium. Magn Reson Med. 1997 Oct;38(4):541-5. doi: 10.1002/mrm.1910380406. PMID 9324319
- [Background] Jerosch-Herold M, Sheridan DC, Kushner JD, Nauman D, Burgess D, Dutton D, Alharethi R, Li D, Hershberger RE. Cardiac magnetic resonance imaging of myocardial contrast uptake and blood flow in patients affected with idiopathic or familial dilated cardiomyopathy. Am J Physiol Heart Circ Physiol. 2008 Sep;295(3):H1234-H1242. doi: 10.1152/ajpheart.00429.2008. Epub 2008 Jul 25. PMID 18660445
- [Background] Pack NA, Dibella EV, Wilson BD, McGann CJ. Quantitative myocardial distribution volume from dynamic contrast-enhanced MRI. Magn Reson Imaging. 2008 May;26(4):532-42. doi: 10.1016/j.mri.2007.10.003. Epub 2008 Feb 20. PMID 18068931
- [Background] Weber KT, Brilla CG. Pathological hypertrophy and cardiac interstitium. Fibrosis and renin-angiotensin-aldosterone system. Circulation. 1991 Jun;83(6):1849-65. doi: 10.1161/01.cir.83.6.1849. PMID 1828192
- [Background] van Hoeven KH, Factor SM. A comparison of the pathological spectrum of hypertensive, diabetic, and hypertensive-diabetic heart disease. Circulation. 1990 Sep;82(3):848-55. doi: 10.1161/01.cir.82.3.848. PMID 2394006
- [Background] Rossi MA. Pathologic fibrosis and connective tissue matrix in left ventricular hypertrophy due to chronic arterial hypertension in humans. J Hypertens. 1998 Jul;16(7):1031-41. doi: 10.1097/00004872-199816070-00018. PMID 9794745
- [Background] McLenachan JM, Dargie HJ. Ventricular arrhythmias in hypertensive left ventricular hypertrophy. Relationship to coronary artery disease, left ventricular dysfunction, and myocardial fibrosis. Am J Hypertens. 1990 Oct;3(10):735-40. doi: 10.1093/ajh/3.10.735. PMID 2145865
- [Background] Beltrami CA, Finato N, Rocco M, Feruglio GA, Puricelli C, Cigola E, Sonnenblick EH, Olivetti G, Anversa P. The cellular basis of dilated cardiomyopathy in humans. J Mol Cell Cardiol. 1995 Jan;27(1):291-305. doi: 10.1016/s0022-2828(08)80028-4. PMID 7760353
- [Background] Anderson KP, Walker R, Urie P, Ershler PR, Lux RL, Karwandee SV. Myocardial electrical propagation in patients with idiopathic dilated cardiomyopathy. J Clin Invest. 1993 Jul;92(1):122-40. doi: 10.1172/JCI116540. PMID 8325977
- [Background] de Bakker JM, van Capelle FJ, Janse MJ, Tasseron S, Vermeulen JT, de Jonge N, Lahpor JR. Fractionated electrograms in dilated cardiomyopathy: origin and relation to abnormal conduction. J Am Coll Cardiol. 1996 Apr;27(5):1071-8. doi: 10.1016/0735-1097(95)00612-5. PMID 8609323
- [Background] Kawara T, Derksen R, de Groot JR, Coronel R, Tasseron S, Linnenbank AC, Hauer RN, Kirkels H, Janse MJ, de Bakker JM. Activation delay after premature stimulation in chronically diseased human myocardium relates to the architecture of interstitial fibrosis. Circulation. 2001 Dec 18;104(25):3069-75. doi: 10.1161/hc5001.100833. PMID 11748102
- [Background] Castillo E, Osman NF, Rosen BD, El-Shehaby I, Pan L, Jerosch-Herold M, Lai S, Bluemke DA, Lima JA. Quantitative assessment of regional myocardial function with MR-tagging in a multi-center study: interobserver and intraobserver agreement of fast strain analysis with Harmonic Phase (HARP) MRI. J Cardiovasc Magn Reson. 2005;7(5):783-91. doi: 10.1080/10976640500295417. PMID 16358393
- [Background] Fernandes VR, Polak JF, Cheng S, Rosen BD, Carvalho B, Nasir K, McClelland R, Hundley G, Pearson G, O'Leary DH, Bluemke DA, Lima JA. Arterial stiffness is associated with regional ventricular systolic and diastolic dysfunction: the Multi-Ethnic Study of Atherosclerosis. Arterioscler Thromb Vasc Biol. 2008 Jan;28(1):194-201. doi: 10.1161/ATVBAHA.107.156950. Epub 2007 Oct 25. PMID 17962621
- [Background] Osman NF, Prince JL. Visualizing myocardial function using HARP MRI. Phys Med Biol. 2000 Jun;45(6):1665-82. doi: 10.1088/0031-9155/45/6/318. PMID 10870717
- [Background] Rosen BD, Saad MF, Shea S, Nasir K, Edvardsen T, Burke G, Jerosch-Herold M, Arnett DK, Lai S, Bluemke DA, Lima JA. Hypertension and smoking are associated with reduced regional left ventricular function in asymptomatic: individuals the Multi-Ethnic Study of Atherosclerosis. J Am Coll Cardiol. 2006 Mar 21;47(6):1150-8. doi: 10.1016/j.jacc.2005.08.078. Epub 2006 Feb 23. PMID 16545644
- [Background] de Simone G, Devereux RB, Koren MJ, Mensah GA, Casale PN, Laragh JH. Midwall left ventricular mechanics. An independent predictor of cardiovascular risk in arterial hypertension. Circulation. 1996 Jan 15;93(2):259-65. doi: 10.1161/01.cir.93.2.259. PMID 8548897
- [Background] Niendorf HP, Haustein J, Cornelius I, Alhassan A, Clauss W. Safety of gadolinium-DTPA: extended clinical experience. Magn Reson Med. 1991 Dec;22(2):222-8; discussion 229-32. doi: 10.1002/mrm.1910220212. PMID 1812350
- [Background] Viollet L, Gailey S, Thornton DJ, Friedman NR, Flanigan KM, Mahan JD, Mendell JR. Utility of cystatin C to monitor renal function in Duchenne muscular dystrophy. Muscle Nerve. 2009 Sep;40(3):438-42. doi: 10.1002/mus.21420. PMID 19623638
- [Background] Nadarajah VD, van Putten M, Chaouch A, Garrood P, Straub V, Lochmuller H, Ginjaar HB, Aartsma-Rus AM, van Ommen GJ, den Dunnen JT, 't Hoen PA. Serum matrix metalloproteinase-9 (MMP-9) as a biomarker for monitoring disease progression in Duchenne muscular dystrophy (DMD). Neuromuscul Disord. 2011 Aug;21(8):569-78. doi: 10.1016/j.nmd.2011.05.011. Epub 2011 Jul 2. PMID 21724396
- [Background] Hollingsworth KG, Garrood P, Eagle M, Bushby K, Straub V. Magnetic resonance imaging in Duchenne muscular dystrophy: longitudinal assessment of natural history over 18 months. Muscle Nerve. 2013 Oct;48(4):586-8. doi: 10.1002/mus.23879. Epub 2013 Aug 30. PMID 23620230
- [Background] Cao Y, Huang DQ, Shih G, Prince MR. Signal Change in the Dentate Nucleus on T1-Weighted MR Images After Multiple Administrations of Gadopentetate Dimeglumine Versus Gadobutrol. AJR Am J Roentgenol. 2016 Feb;206(2):414-9. doi: 10.2214/AJR.15.15327. Epub 2015 Dec 23. PMID 26700156
- [Background] Jost G, Lenhard DC, Sieber MA, Lohrke J, Frenzel T, Pietsch H. Signal Increase on Unenhanced T1-Weighted Images in the Rat Brain After Repeated, Extended Doses of Gadolinium-Based Contrast Agents: Comparison of Linear and Macrocyclic Agents. Invest Radiol. 2016 Feb;51(2):83-9. doi: 10.1097/RLI.0000000000000242. PMID 26606548